CLINICAL TRIAL: NCT05571800
Title: The Effects of Fresh Mango Consumption in Indices of Glycemic Control, Cardiovascular Health, and Body Composition in Normal Weight, Overweight and Obese Individuals with Prediabetes
Brief Title: Effect of Mango Consumption on Individuals with Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Mango Board (Other)
Responsible Party: Principal Investigator, Hickner, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00002545
Record Dates: First submitted 2022-09-06; First posted 2022-10-07 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: PreDiabetes; Obesity
Keywords: Glycemic Control; Cardiovascular Health; Overweight; Obese; Glycemic Indices; Body Composition
MeSH Terms: conditions — Prediabetic State; Obesity; Overweight | interventions — Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: Randomized, calorie-match controlled
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mango Supplement (Experimental): Participants will consume 120g of fresh mango per day for 24 weeks
  Interventions: Other: Mango
- Placebo Matched Supplement (Placebo Comparator): Participants will consume 200g isocaloric granola bar per day for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Mango — 120g of fresh Mango
  Arms: Mango Supplement
Other: Placebo — 200g isocaloric Granola Bar
  Arms: Placebo Matched Supplement

SUMMARY:
This study is designed to explore the effect of mango consumption on glycemic indices, cardiovascular health, and body composition in overweight and obese individuals with prediabetes.

DETAILED DESCRIPTION:
According to the Centers for Disease Control and Prevention (2016), at least 100 million adults in the United States are diagnosed as pre-diabetic or Type 2 diabetic. With the number of cases steadily increasing in this population, healthcare costs have subsequently increased for both the patient and the health care system. To date, there are few studies (limited to animal model and obese Type 2 diabetic humans) that have examined the efficacy of mangoes on health outcomes, particularly related to diabetes. Therefore, the purpose of the current study is to examine the effect of fresh mango on glycemic indices, body composition, and vascular health measures. Upon favorable outcomes, and with more definite evidence from human studies, mangoes can potentially be implemented in America's diet to help mitigate the advancement and diagnoses of pre and Type 2 diabetes and, as a result, aid in a reduction of healthcare costs. The current study is a 24- week, randomized, controlled experiment including 40 overweight or obese, pre-diabetic men and post-menopausal women aged 50 to 70 years with no diagnosed cardiovascular, metabolic, kidney, or other types of chronic disease to be included. Participants will be randomly assigned to one of two groups: 1) one fresh Tommy Atkins mango (120 g) per day or 2) an isocaloric granola bar per day for 24 weeks. Visits will include anthropometric measurements, glucose, and A1C values via finger prick, venous blood samples to analyze biomarkers related to glycemic control and lipid profiles, vascular measures, and body composition. To analyze the effects of the treatment, ANOVA and Bonferroni's test will be utilized. The investigators hypothesize that daily consumption of one mango per day for 24 weeks will improve the indices of glycemic control, cardiovascular health, and body composition in overweight and obese individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Free of any chronic diseases such as cancer
* BMI of 18.5 kg/m2 to 34.9 kg/m2
* wHbA1c values are 100 mg/dl to 125 mg/dl and HbA1C of 5.7-6.4 %

Exclusion Criteria:

* Individuals diagnosed with cardiovascular diseases (CVD), type 2-diabetes, type 1 diabetes mellitus, other active chronic diseases such as cancer, asthma, glaucoma, kidney, liver and pancreatic disease
* Uncontrolled hypertension (≥160/100 mmHg)
* BMI <18.5 kg/m2 or >34.9 kg/m2
* Not post-menopausal or have been taking hormone replacement therapy for less than 3 months
* taking more than one anti-hypertensive or have been taking them for less than 3 months
* Participating in a weight loss program or having lost or gain ≥10% bodyweight within the last 6 months
* Smoke more than 1 pack/day
* Consumption of >12 alcoholic drinks/week
* Frequent mango consumers (>5 servings/2weeks)
* In concurrent participation with another investigational study
* Currently consuming any performance supplement (i.e. creatine, nitric oxide, whey/casein protein, branched chain amino acids).

  * None of the following special populations will be included: adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, or prisoners.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Effect of mango consumption on glycemic control using blood glucose measures | 3 years
  Blood glucose measures evaluated with finger prick and blood glucose meter
Effect of mango consumption on glycemic control using HbA1c | 3 years
  HbA1c evaluated by finger prick and DCA analyzer
Effect of mango consumption on glycemic control evaluated by Insulin | 3 years
  Insulin evaluated by blood draw Enzyme-linked immunosorbent assay
Effect of mango consumption on glycemic control evaluated by HOMA-IR | 3 years
  HOMA-IR evaluated by blood draw 20 ml Enzyme-linked immunosorbent assay
Effect of mango consumption on glycemic control evaluated by HOMA-β | 3 years
  HOMA-β evaluated by blood draw 20 ml and Enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Effect of mango consumption on indicators of cardiovascular health evaluated by systolic and diastolic blood pressure | 3 years
  Systolic and diastolic blood pressure evaluated by automated blood pressure monitor
Effect of mango consumption on indicators of cardiovascular health evaluated by Indirect bioassay of in vivo endothelial function with FMD | 3 years
  Flow-mediated dilation (FMD) evaluated with high-resolution doppler ultrasound (HD11XE, Phillips Ultrasound, Bothwell, WA, USA) with a 3-12 MHz linear array transducer
Effect of mango consumption on indicators of cardiovascular health evaluated by Indirect bioassay of in vivo endothelial function with PWV | 3 years
  Pulse wave velocity (PWV) evaluated with Sphygmocor for pulse wave velocity, aortic blood pressure and augmentation index
Effect of mango consumption on indicators of cardiovascular health evaluated by Indirect bioassay of in vivo endothelial function with ET-1 | 3 years
  Endothelin-1 (ET-1) evaluated with Enzyme-linked immunosorbent assay
Effect of mango consumption on indicators of cardiovascular health evaluated by biomarker of inflammation (C-reactive protein) | 3 years
  biomarker of inflammation (C-reactive protein) evaluated by blood draw 20 ml and enzyme-linked immunosorbent assay
Effect of mango consumption on indicators of cardiovascular health evaluated by lipid profile | 3 years
  lipid profile evaluated by blood draw and enzyme-linked immunosorbent assay consisting of
  * Triglycerides (TG)
  * Total cholesterol (TC)
  * Low-density lipoprotein cholesterol (LDL-C)
  * Oxidized LDL (Ox-LDL)
  * High-density lipoprotein cholesterol (HDL-C)
Atherogenic risk ratio (TC/HDL-C, LDLC/HDL-C, HDL-C/LDL-C) | 3 years
  Effect of mango consumption on indicators of cardiovascular health evaluated by lipid profile
Effect of mango consumption on body composition evaluated by lean mass | 3 years
  Lean mass evaluated by bioimpedance spectroscopy (BIS)
Effect of mango consumption on body composition evaluated by fat mass | 3 years
  fat mass evaluated by bioimpedance spectroscopy (BIS)
Effect of mango consumption on body composition evaluated by phase angle (PA) | 3 years
  Phase angle (PA) calculated directly from reactance and resistance using the following formula: PA=arctangent reactance(ohm)/resistance (ohm) ×180°/π
Effect of mango consumption on body composition evaluated by weight | 3 years
  Weight evaluated by Ohaus Portable Electronic CS Series Scales
Effect of mango consumption on anthropometric measure of Waist circumference (WC) | 3 years
  evaluated by Gulick fiberglass measuring tape with a tension handle
Effect of mango consumption on anthropometric measure of HC | 3 years
  hip circumference (HC) evaluated by Gulick fiberglass measuring tape with a tension handle
Effect of mango consumption on anthropometric measure WC/HC ratio | 3 years
  waist to hip ratio (WC/HC)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hickner, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States